CLINICAL TRIAL: NCT06659562
Title: Phase Ib Safety, Tolerability and Pharmacokinetic Study of Subcutaneously Administered HER-096 in Healthy Volunteer Subjects and Patients With Parkinson's Disease
Brief Title: Clinical Study of HER-096 in Healthy Volunteer Subjects and Patients With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herantis Pharma Plc. (Industry)
Collaborators: Clinical Research Services Turku - CRST Ltd (Unknown); BC Platforms (Unknown); Oy Medfiles Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-XC-CL; 2024-512532-30-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-11; First posted 2024-10-26 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: HER-096; Safety and Tolerability Study; Healthy Volunteer Subjects; PD; Parkinson Disease; Central Nervous System Disorders; Neurodegenerative Disorders
MeSH Terms: conditions — Parkinson Disease; Central Nervous System Diseases; Neurodegenerative Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Part 1: Single dose cohort in older and elderly (50-75 years of age) healthy volunteer subjects.
  Part 2: Two multiple dose cohorts in patients with mild or moderate PD (45-80 years of age).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1: Open-label. Part 2: Double-blind, randomized, placebo-controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HER-096 (Part 1) (Active Comparator): Older and elderly healthy volunteer subjects
  Interventions: Drug: HER-096
- HER-096 (Part 2) (Active Comparator): Parkinson's Disease patients
  Interventions: Drug: HER-096
- Placebo (Part 2) (Placebo Comparator): Parkinson's Disease patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HER-096 — Administered as a single dose via s.c. injection
  Arms: HER-096 (Part 1)
Drug: HER-096 — Administered as multiple doses via s.c. injection. Administered twice a week (2 doses/week) during a 4-week period.
  Arms: HER-096 (Part 2)
Drug: Placebo — Administered as multiple doses via s.c. injection. Administered twice a week (2 doses/week) during a 4-week period.
  Other Names: Sodium chloride 9 mg/ml; 0.9% physiological saline solution
  Arms: Placebo (Part 2)

SUMMARY:
In this clinical study, the safety and tolerability of HER-096 and the way the body interacts with the drug (pharmacokinetics) will be investigated. The clinical study consists of two parts. In Part 1, the drug HER-096 is given as a single dose to healthy volunteer subjects. In Part 2, HER-096 or placebo (physiological saline) is given as multiple doses during a 4-week period to patients with Parkinson´s disease. The doses are given as injections under the skin (subcutaneous injection).

DETAILED DESCRIPTION:
This is a Phase Ib clinical study, in which safety, tolerability and pharmacokinetic profile of HER-096 will be investigated after a subcutaneously (s.c.) administered single dose in healthy volunteer subjects (HVS) in an open-labelled Part 1 and after multiple s.c. administered doses in patients with Parkinson´s disease (PD) in a randomised, placebo-controlled Part 2. In Part 2, two out of three patients will receive active HER-096 treatment and one out of three patients will receive a placebo solution. Novel biomarkers related to the treatment will be explored.

The total study duration per subject is approximately 50 days in Part 1 and 100 days in Part 2 consisting of screening, treatment and safety follow-up periods. In total, 8-12 male or female HVS and 24-28 male or female PD patients will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

1. Sufficient command of the Finnish language to be able to understand the subject information leaflet and to communicate well with the study personnel.
2. Age 50-75 years at the time of consent.
3. Male or postmenopausal female.
4. BMI 18-35 kg/m2
5. Good general health, based on medical history, physical examination and laboratory assessments.
6. Provision of written informed consent prior to any other trial related procedure is performed.
7. Judged by the investigator to be alert and oriented to person, place, time and situation when giving the informed consent.

Part 2:

1. Provision of written informed consent prior to any other trial related procedure is performed.
2. Clinically established diagnosis of PD (MDS 2015 criteria), early idiopathic, Modified Hoehn and Yahr scale up to 2.5, with bradykinesia plus one of the other cardinal signs of PD (resting tremor, rigidity) being present, without any other known or suspected cause of PD.
3. Brain DAT-SPECT or DAT-PET imaging results consistent with PD.
4. Age 45-80 years at the time of consent; males and postmenopausal females.
5. Stable clinical disease state with either:

   1. Patient does not require dopaminergic PD medication and is not expected to require dopaminergic treatment within the study duration, or
   2. Stable treatment including one or any combination of below treatments, as clinically established and well tolerated

   i. Levodopa substitution with oral levodopa + DOPA decarboxylase inhibitor (not more than 1000 mg levodopa daily) ii. Orally administered dopamine agonists excluding ergot-derived- agonist drugs iii. Transdermal rotigotine patches iv. Monoamine oxidase B (MAO-B) inhibitor c. All treatments of PD should be stable for at least 45 days prior to baseline assessments and not expected to change within the study duration.
6. Good general health (apart from PD), based on medical history, physical examination and laboratory assessments.
7. BMI 18-35 kg/m2.

Exclusion Criteria:

Part 1:

1. Predicted poor compliance with study procedures, restrictions and requirements.
2. Veins unsuitable for repeated venepuncture or cannulation.
3. History or evidence of current clinically significant cardiovascular, pulmonary, renal, hepatic, gastrointestinal, haematological, metabolic-endocrine, neurological, urogenital or psychiatric disorder. Subjects with any type of generalized seizures in adulthood must be excluded. Personal or first-degree family history of congenital long QT syndrome or sudden death of a first-degree relative suspected to be due to long QT syndrome will also exclude the subject.
4. MRI (3 T) of the brain with indication of clinically significant CNS disorder.
5. History of any type of cancer, except for the age group of above 65 years, where a history of successfully treated cancer, with at least 5 years since the end of treatment, or local prostate cancer with no evidence of disease progression under adequate active surveillance, may be allowed at the investigator's discretion.
6. Susceptibility to severe allergic reactions, e.g. history of anaphylactic shock due to any reason.
7. Any condition requiring regular concomitant medication (including non-prescriptional over-the-counter (OTC) drugs), or likely to need any concomitant medication during the study. As exceptions, hormone replacement therapy in female subjects and supplementation therapy with thyroxin, iron, calcium, folate and vitamin B12 at recommended doses is allowed. Vitamin D supplementation at doses of 20 µg/day or less is also allowed. The use of other vitamins, nutritional supplements and herbal products, at recommended doses, may be allowed at the investigator's discretion. Occasional use of paracetamol for pain is allowed.
8. Use of any medication that might affect the study results or cause a health risk for the subject within 2 weeks prior to IMP administration.
9. Any clinically significant abnormalities in screening laboratory test results, vital signs or physical examination findings that might influence the results of the study or cause a health risk for the subject if he/she takes part in the study.
10. Estimated glomerular filtration rate (eGFR) below 60 ml/min/1,73 m2
11. Coagulopathy, thrombocytopenia, use of anticoagulants or other antithrombotic agents.
12. Positive serology to human immunodeficiency virus antibodies (HIVAgAb), hepatitis C virus antibodies (HCVAb) or hepatitis B surface antigen (HBsAg).
13. Any clinically significant 12-lead ECG abnormality after 10 min rest in supine position at the screening visit or baseline evaluation at the dosing visit. For example, any of the following findings in the resting ECG:

    1. QTcF above 450 or below 300 msec;
    2. Notable resting bradycardia (heart rate (HR) below 45 beats per minute (bpm)) or tachycardia (HR above 100 bpm);
    3. Screening or baseline ECG with QRS and/or T wave judged to be unfavourable for a consistently accurate QT measurement (e.g., neuromuscular artifact that cannot be readily eliminated, arrhythmias, indistinct QRS onset, low amplitude T wave, merged T- and U-waves, prominent U waves);
    4. Evidence of atrial fibrillation, atrial flutter, complete bundle branch block, Wolf-Parkinson-White syndrome, or cardiac pacemaker.
14. HR below 45 bpm or above 85 bpm, systolic blood pressure (BP) below 90 mmHg or above 150 mmHg, or diastolic BP below 50 mmHg or above 95 mmHg after 10 min rest in supine position at the screening visit.
15. History of alcohol or drug abuse within the last 5 years, or current regular use of illicit drugs or excessive use of alcohol (regular alcohol drinking of more than 24 units/week for males or 14 units/week for females).
16. Positive breath test for alcohol or positive urine screening test result for drugs of abuse.
17. Current use of nicotine-containing products of more than 5 cigarettes or equivalent per day, or inability to refrain from using nicotine-containing products during the stay at the study centre.
18. Inability to refrain from consuming caffeine-containing beverages during the stay at the study centre.
19. Participation in any other clinical drug study within 3 months before the IMP administration of this study.
20. Donation of blood within 3 months before the IMP administration.
21. Any medical or surgical procedure planned during the study period.
22. Male subjects who are sexually active with a female partner of childbearing potential and do not agree to use two medically accepted methods of contraception during the study and for three months after the dosing, and refrain from donating sperm during this time.
23. Female subjects need to be postmenopausal for at least one (1) year before participation or be surgically sterilized.
24. Any indication of increased intracerebral pressure by neurological examination or other contraindication for lumbar puncture.
25. Any contraindication for MRI of the brain.
26. Large tattoo or another condition of the skin or subcutaneous tissue that would prevent reliable assessment of local injection site reactions.
27. Significant risk of suicidal behaviour, defined using the C-SSRS, as the subject answering "yes" at the screening visit to suicidal ideation questions 4 or 5 or answering "yes" to suicidal behaviour within the past 6 months.

Part 2:

1. Predicted poor compliance with study procedures, restrictions and requirements.
2. Veins unsuitable for repeated venepuncture or cannulation.
3. History or evidence of current clinically significant, potentially unstable cardiovascular, pulmonary, renal, hepatic, gastrointestinal, haematological, metabolic-endocrine or urogenital disorder. Persons with stable chronic diseases may be included at the investigator's discretion. Subjects with any type of generalized seizures in adulthood must be excluded. Personal or first-degree family history of congenital long QT syndrome or sudden death of a first-degree relative suspected to be due to long QT syndrome will also exclude the subject.
4. History of major psychiatric disorder, including schizophrenia and bipolar illness. A subject with a history of major depressive disorder (MDD) that is considered to be in remission or controlled with treatment can be included in the trial per investigator's judgement.
5. History of any type of cancer, except for the age group of above 65 years, where a history of successfully treated cancer, with at least 5 years since the end of treatment, or local prostate cancer or fully excised non-melanoma skin cancers with no evidence of disease progression under adequate active surveillance for at least 6 months, or cervical intraepithelial neoplasia stage I uterine cancer may be allowed at the investigator's discretion.
6. Other neurological disorder than PD, including Alzheimer's disease, ALS, multiple sclerosis, corticobasal degeneration (CBD), progressive supranuclear palsy (PSP), multiple system atrophy (MSA), Parkinson's disease dementia (PDD) and other movement disorders with overlapping symptomatology to PD.
7. Wearing-off or dyskinesia in relation to dopaminergic treatment.
8. Treatment with levodopa infusions, apomorphine infusions or other non-oral PD medications (except for transdermal rotigotine patches).
9. Ongoing or previous treatment of PD with deep brain stimulation (DBS) or high-intensity ultrasound (HIFU).
10. Coagulopathy, thrombocytopenia, use of anticoagulants or other antithrombotic agents.
11. Susceptibility to severe allergic reactions, e.g. history of anaphylactic shock due to any reason.
12. Ongoing treatment with antipsychotic medications, or use of other medications that in the opinion of the investigator might cause a risk for the study participant or jeopardise the study assessments. Disallowed medications include e.g. systemically used glucocorticoids and other modulators of immune functions.
13. Any clinically significant abnormalities in screening laboratory test results, vital signs or physical examination findings that might influence the results of the study or cause a health risk for the subject if he/she takes part in the study.
14. Estimated glomerular filtration rate (eGFR) below 60 ml/min/1,73 m2
15. Positive serology to human immunodeficiency virus antibodies (HIVAgAb), hepatitis C virus antibodies (HCVAb) or hepatitis B surface antigen (HBsAg).
16. History of alcohol or drug abuse within the last 5 years, or current regular use of illicit drugs or excessive use of alcohol (regular alcohol drinking of more than 24 units/week for males or 14 units/week for females).
17. Positive breath test for alcohol or positive urine screening test result for drugs of abuse.
18. Current use of nicotine-containing products of more than 10 cigarettes or equivalent per day, or inability to refrain from using nicotine-containing products during the stay at the study centre.
19. Participation in any other clinical drug study within 3 months before the first IMP administration of this study.
20. Donation of blood within 3 months before the first IMP administration.
21. Any medical or surgical procedure planned during the study period.
22. Male subjects who are sexually active with a female partner of childbearing potential and do not agree to use two medically accepted methods of contraception during the study and for three months after the last dosing, and refrain from donating sperm during this time.
23. Female subjects need to be postmenopausal for at least one (1) year before participation or be surgically sterilized.
24. Any contraindication MRI of the brain.
25. MRI (3 T) of the brain with indication of clinically significant CNS disorder apart from PD.
26. For subjects scheduled to undergo DAT-SPECT: any contraindication for DAT-SPECT of the brain, including previous hypersensitivity reactions to iodine administration.
27. Any indication of increased intracerebral pressure by neurological examination at inclusion, or another contraindication for LP.
28. Any condition expected to require changes in medical treatment during the trial period, or use of disallowed concomitant medications, or concomitant medication that has not been stable for at least 45 days prior to baseline assessments. The use vitamins, nutritional supplements and herbal products, at recommended doses, may be allowed at the investigator's discretion. Occasional use of paracetamol for pain is allowed. Hormone replacement therapy in female subjects and supplementation therapy with thyroxin, iron, calcium, folate and vitamin B12 at recommended doses is allowed. Vitamin D supplementation at doses of 20 µg/day or less is also allowed.
29. Large tattoo or another condition of the skin or subcutaneous tissue that would prevent reliable assessment of local injection site reactions.
30. Significant risk of suicidal behaviour, defined using the C-SSRS, as the subject answering "yes" at the screening visit to suicidal ideation questions 4 or 5 or answering "yes" to suicidal behaviour within the past 6 months.
31. Previous treatment with any investigational and/or marketed passive immunotherapy against PD within 6 months before screening or 5 half-lives, whichever is longer, unless there is firm evidence that the subject received placebo only (in the case of any investigational product administered within the frame of a clinical trial participation).
32. Participation in previous clinical trials for PD and/or for neurological disorders using any small molecule drug with a washout <30 days or <5 half-lives of the drug, whichever is longer before screening, unless there is firm evidence that the subject received placebo only.
33. Concomitant participation in any other clinical trial using experimental or approved medications or therapies (e.g., device, stem cells). This does not include noninterventional devices for disease tracking or imaging studies.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events (TEAEs) | From start of treatment (Day 0) to end of study (Day 8, Part 1 and Day 52, Part 2).
  Incidence, type and severity of TEAEs
Physical Examination | From start of treatment (Day 0) to end of study (Day 8, Part 1 and Day 52, Part 2).
  Incidence of clinically significant physical examination findings
Vital Signs | From start of treatment (Day 0) to end of study (Day 8, Part 1 and Day 52, Part 2).
  Incidence of clinically significant findings in systolic and diastolic blood pressure, heart rate and body temperature
Laboratory safety assessments - Haematology | From start of treatment (Day 0) to end of study (Day 8, Part 1 and Day 52, Part 2).
  Incidence of clinically significant laboratory variables in haemoglobin, erythrocytes, leucocytes, thrombocytes, mean corpuscular volume (MCV), mean corpuscular haemoglobin concentration (MCHC) and differential leucocyte count
Laboratory safety assessments - Clinical chemistry | From start of treatment (Day 0) to end of study (Day 8, Part 1 and Day 52, Part 2).
  Incidence of clinically significant laboratory variables in alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT), bilirubin total, bilirubin conjugated, albumin, creatinine, glucose, sodium, potassium, calcium, C-reactive protein (CRP), creatine kinase (CK), thyroid-stimulating hormone (TSH), estimated glomerular filtration rate (eGFR) and prolactin.
Laboratory safety assessments - Coagulation | From start of treatment (Day 0) to end of study (Day 8, Part 1 and Day 52, Part 2).
  Incidence of clinically significant laboratory variables in plasma activated partial thromboplastin time (P-APTT) and international normalized ratio (INR)
Laboratory safety assessments - Urinalysis | From start of treatment (Day 0) to end of study (Day 8, Part 1 and Day 52, Part 2).
  Incidence of clinically significant laboratory variables in pH, erythrocytes, leukocytes, nitrite, protein, glucose, ketones and urine creatinine
12-lead electrocardiogram (ECG) | From start of treatment (Day 0) to Day 2 in Part 1, and Day 52 in Part 2.
  Incidence of clinically significant findings in heart rate, PR interval, RR, QRS interval and QTcF
Magnetic Resonance Imaging (MRI) of the brain | From start of treatment (Day 0) to Day 52
  Number of participants with new brain microhaemorrhages (microbleeds) as assessed with MRI of the brain in Part 2
Columbia-Suicide Severity Rating Scale (C-SSRS) | From start of treatment (Day 0) to end of study (Day 8 in Part 1 and Day 52 in Part 2).
  Incidence of subjects with increased suicidal tendencies measured by C-SSRS questionnaire consisting of maximum of 4 sections.
  Suicidal ideation: 5 yes/no questions with ´YES´ indicating suicidal ideation and ´NO´ indicating no suicidal ideation.
  Intensity of ideation: 5 questions to be rated with respect to the most severe type if ideation (5 being the most severe intensity and 1 being the least intensity).
  Suicidal behavior: 5 yes/no questions with ´YES´ indicating suicidal behavior and ´NO´ indicating no suicidal behavior.
  Actual attempts only: 2 questions to be rated with respect to the most severe outcome of the suicide attempt (highest score indicating the most severe outcome and 0 indicating no harm).
Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I-III | Day 1 to Day 52
  Score changes in MDS-UPDRS.
  Part I: non-motor experiences of daily living
  Part II: motor experiences of daily living
  Part III: motor examinations
  Questions are answered on a scale 0-4, 0 being considered as a normal state and 4 as a severe state. The highest total score of Parts I-III is 180 points.
  Applicable in Part 2 of the study only.

SECONDARY OUTCOMES:
HER-096 concentration levels in plasma and urine | 24 hours
  Changes in HER-096 concentration levels in plasma and urine
HER-096 concentration in CSF | Up to 72 hours
  Changes in HER-096 concentration levels in CSF.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Juha Rinne, MD, PhD, Principal Investigator — Clinical Research Services Turku - CRST Oy
Locations (1):
- Clinical Research Services Turku - CRST Oy, Turku, Finland, Finland